CLINICAL TRIAL: NCT05781841
Title: Assessment Of Gene Expression Of Suppressor Of Cytokine 3, Interferons Alpha And Beta In Cutaneous Warts
Brief Title: Gene Expression Of Suppressor Of Cytokines in In Cutaneous Warts
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reham Helal Aboelhamd, principal investigator, Sohag University
Other Study IDs: Soh-Med-23-03-7MS
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Warts
Keywords: HPV; Warts; STAT1; SOCS 3
MeSH Terms: conditions — Warts

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Under complete sterile precautions, Skin biopsy will be taken from healthy volunteers of the control group via 2 mm disposable punches and from patients with wart lesion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with cutaneous warts: Under complete sterile precautions, Skin biopsy will be taken from patients with wart lesion.
  The specimen will be put in sterile plane tube containing saline and will be transferred immediately to the central research laboratory to be processed
  Interventions: Diagnostic Test: Detection of expression of SOCS3 gene; Diagnostic Test: Detection of expression of IFN-α gene; Diagnostic Test: Detection of expression of IFN-β gene
- healthy volunteers: Under complete sterile precautions, Skin biopsy will be taken from healthy volunteers of the control group via 2 mm disposable punches .
  The specimen will be put in sterile plane tube containing saline and will be transferred immediately to the central research laboratory to be processed
  Interventions: Diagnostic Test: Detection of expression of SOCS3 gene; Diagnostic Test: Detection of expression of IFN-α gene; Diagnostic Test: Detection of expression of IFN-β gene

INTERVENTIONS:
Diagnostic Test: Detection of expression of SOCS3 gene — Detection of expression of SOCS3, in each samples using Real-Time PCR
Diagnostic Test: Detection of expression of IFN-α gene — Detection of expression of IFN-α gene in each samples using Real-Time PCR
Diagnostic Test: Detection of expression of IFN-β gene — Detection of expression of IFN-β gene in each samples using Real-Time PCR

SUMMARY:
Warts are common epidermal growths caused by various strains of human papilloma virus (HPV). Viral warts are common with a prevalence rate of 7-12%.

Human papilloma virus is small non enveloped viruses that contain a double-stranded DNA genome. There are more than 200 HPV genotypes are reported, however, the high-risk types, including HPV genotype-16 (HPV16), 18, 31, and 45, are the causes of 80% of cervical cancers.

DETAILED DESCRIPTION:
Cutaneous warts are benign lesions caused by low risk-HPV. Of which the most prevalent genotypes are HPV1/2/3/4/10/27/57, and from these genotypes 1, 2, 4, 27, 57 cause common warts. Palmoplantar warts can be caused by genotypes 1 and 2. Condyloma acuminata (anogenital warts) are common sexually transmitted infections caused primarily by HPV-6 and HPV-11 (in 90% of cases) and occasionally by HPV-16 and HPV-18.

About 90% of HPV infections are eliminated within two years due to an efficient immune response. In the form of correct activation of the elements of the innate immune response, such as macrophages, polymorphonuclear cells, natural killer (NK) cells, which release immunomodulatory molecules that help control the infection. In addition, HPV-infected keratinocytes may act as non-professional antigen-presenting cells to promote the clearance of infected cells through the secretion of antiviral and pro-inflammatory mediators.

Interferon (IFN) belongs to a family of inducible cytokines which promote an"antiviral state" in infected cells and neighboring cells through the activation of interferon-stimulated genes (ISG). Three IFN types have been identified (type I, II and III), of which I and III are involved in the innate immune response. Type I IFNs include IFN-α, IFN-β, IFN-ɛ, IFN-κ and IFN-ω.

Most type I IFNs are induced through the binding of viral products to pattern recognition receptors, leading to activation of interferon response factors to drive the synthesis of IFN molecules. After secretion, type I IFNs bind to its receptor, which induces the phosphorylation of signal transducer and activator of transcription 1 (STAT1) and STAT2, which then translocate to the nucleus to induce transcription of (ISGs).

The antiviral effects of IFN-I are mediated by inducing several (ISGs) which impair viral replication through inhibition of protein translation and degradation of viral RNA. ISGs also activate the survival of innate and adaptive immune cells including dendritic cells, macrophages, NK cells and T cells. So, IFN-I helps to control the infections.

During the viral infection process, cytokines trigger and deal with inflammation. However, excessive production of cytokines can cause a cytokine storm, and excessive host innate immune response can also damage the body. Therefore, the suppressor of cytokine signaling proteins with negative feedback regulation ability, prevents the excessive secretion of cytokines from harming the host cell. These intracellular protein family is constituted by suppressor of cytokine signaling proteins 1-7, Which are potent endogenous inhibitors of Janus kinase (JAK/ STAT) signal.

The SOCS 3 is mainly involved in the negative feedback regulation of the tyrosine-protein kinase/ STAT signaling. The critical role of SOCS3 is manifested by its binding to both the JAK and the tyrosine kinase receptor, which further inhibits STAT3 phosphorylation. The JAK/STAT pathway transduces extracellular signals to the nucleus. Its activation stimulates cell proliferation, differentiation, migration, and immune challenge. The JAK/STAT signaling pathway plays an important role in viral infection.

The SOCS family are induced by various viral infections, including human immunodeficiency virus-1, hepatitis B and C viruses, herpes simplex virus type 1, respiratory syncytial virus, Ebola virus, influenza A, and coxsackie virus. Influenza A virus inhibits type I IFN signaling through the induction of SOCS3 expression. Newcastle disease virus (NDV) infection activates the expression of SOCS3 at the mRNA and protein level, which is conducive to the virus replication.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with cutaneous warts of various types aged 18-50 years old.

Exclusion Criteria:

* 1. Pregnancy 2. Lactation 3. Patient on anti-inflammatory and antioxidant drugs 4. Skin infections, other than warts 5. Skin diseases 6. Systemic infection. 7. Malignancies

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: A-patients: - The study will include 35 patients with cutaneous warts aged18-50 years old and 15 age matched controls (blood donors).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
This study aims to assess the expression of genes of SOCS3 in cutaneous warts. | from april 2023 to December 2023
  Under complete sterile precautions, Skin biopsy will be taken from healthy volunteers of the control group via 2 mm disposable punches and from patients with wart lesion.
  The specimen will be put in sterile plane tube containing saline and will be transferred immediately to the central research laboratory to be processed as follow:
  1. Tissue grinding into smaller pieces then will be subjected for RNA extraction by automated kits according to its manufacture instruction.
  2. Conversion of RNA to double stranded DNA using RT( reverse transcriptase conversion Kits ) according to its manufacture instruction using conventional PCR.
  3. Detection of expression of SOCS3 gene in each samples using Real-Time PCR
This study aims to assess the expression of genes of IFN-α in cutaneous warts. | from April 2023 to December 2023
  Under complete sterile precautions, Skin biopsy will be taken from healthy volunteers of the control group via 2 mm disposable punches and from patients with wart lesion.
  The specimen will be put in sterile plane tube containing saline and will be transferred immediately to the central research laboratory to be processed as follow:
  1. Tissue grinding into smaller pieces then will be subjected for RNA extraction by automated kits according to its manufacture instruction.
  2. Conversion of RNA to double stranded DNA using RT( reverse transcriptase conversion Kits ) according to its manufacture instruction using conventional PCR.
  3. Detection of expression of IFN-α gene in each samples using Real-Time PCR
This study aims to assess the expression of genes of IFN-β in cutaneous warts. | from April 2023 to December 2023
  Under complete sterile precautions, Skin biopsy will be taken from healthy volunteers of the control group via 2 mm disposable punches and from patients with wart lesion.
  The specimen will be put in sterile plane tube containing saline and will be transferred immediately to the central research laboratory to be processed as follow:
  1. Tissue grinding into smaller pieces then will be subjected for RNA extraction by automated kits according to its manufacture instruction.
  2. Conversion of RNA to double stranded DNA using RT( reverse transcriptase conversion Kits ) according to its manufacture instruction using conventional PCR.
  3. Detection of expression of IFN-β gene in each samples using Real-Time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Hanan A Assaf, professor, Study Chair — Sohag University; Zeinab A Goda, lecturer, Study Chair — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feng M, Xie T, Li Y, Zhang N, Lu Q, Zhou Y, Shi M, Sun J, Zhang X. A balanced game: chicken macrophage response to ALV-J infection. Vet Res. 2019 Mar 6;50(1):20. doi: 10.1186/s13567-019-0638-y. PMID 30841905
- See also: Related Info — http://doi.org/10.3389/fcimb.2021.748795